CLINICAL TRIAL: NCT00075829
Title: A Trial of Tandem Autologous Stem Cell Transplants +/- Post Second Autologous Transplant Maintenance Therapy vs Single Autologous Stem Cell Transplant Followed by Matched Sibling Non-myeloablative Allogeneic Stem Cell Transplant for Patients With Multiple Myeloma (BMT CTN #0102)
Brief Title: Stem Cell Transplantation in Individuals With Multiple Myeloma (BMT CTN 0102)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0102; BMT CTN 0102 (Other: Blood and Marrow Transplant Clinicial Trials Network); SUMC-79730 (Other: Institutional Review Board at SUMC); 417 (Other: NHLBI); NCT00321607 (obsolete NCT alias); NCT00386568 (obsolete NCT alias)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma
Keywords: Stage II Multiple Myeloma; Stage III Multiple Myeloma; Refractory Plasma Cell Neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Dexamethasone; Calcium Dobesilate; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auto transplants plus Therapy (Active Comparator): One autologous transplant along with a second autologous transplant will be preformed followed by one year of Dexamethasone and Thalidomide maintenance therapy.
  Interventions: Procedure: One Autologous Transplant; Procedure: Second Autologous Transplant; Drug: Thalidomide; Drug: Dexamethasone
- Auto transplants (Active Comparator): One autologous transplant along with a second autologous transplant will be preformed followed by one year of observation.
  Interventions: Procedure: One Autologous Transplant; Procedure: Second Autologous Transplant; Behavioral: Observation
- Auto and Allo transplants (Active Comparator): One autologous transplant and one non-myeloablative allogeneic transplant will be preformed and followed by one year of observation.
  Interventions: Procedure: One Autologous Transplant; Procedure: Non-Myeloablative Allogeneic Transplant; Behavioral: Observation

INTERVENTIONS:
Procedure: One Autologous Transplant — Melphalan will be administered at a dose of 200 mg/m2. Melphalan will be given in one dose infused on Day -2. Melphalan dose is based on ideal body weight (IBW) for patients who weigh 100-120% of their IBW. All patients will receive an autologous graft with a minimum cell dose of 2.0 x 106 CD34+ cells/kg patient weight. Patients will receive ~5 ug/kg/day of Granulocyte-Colony Stimulating Factor (G-CSF) subcutaneously from Day 5 post-transplant until absolute neutrophil count (ANC) > 500/mm3 for two days.
Procedure: Non-Myeloablative Allogeneic Transplant — Upon recovery and at least Day 60 post-autograft, patients with an available 6/6 HLA matched sibling will receive an allograft after non-myeloablative conditioning. Day 0 patients will receive Total Body Irradiation (TBI) 2.0 Gy from a linear accelerator ≤ 20 cGy/min, followed by allogeneic peripheral blood stem cell (PBSC) infusion. Commence cyclosporine (CSA) on Day -3 at 5 mg/kg bid PO for a daily dose of 10 mg/kg/day through Day +84 based on actual body weight. Starting on Day 84, patients in partial or complete response with the absence of graph versus host disease (GVHD) will have CSA tapered so the patient will be off CSA by Day 180. Oral administration of Mycophenolate Mofetil will be at a daily dose of 30 mg/kg/day from the evening of Day 0 until Day 27 post-transplant.
  Arms: Auto and Allo transplants
Procedure: Second Autologous Transplant — Upon recovery from the first autograft, but at least 60 days (preferably between 60-120 days) after the first autograft, patients without an HLA-matched sibling donor will receive a second autograft, also conditioned with melphalan 200 mg/m2.
  Arms: Auto transplants; Auto transplants plus Therapy
Drug: Thalidomide — Patients will be initiated on a starting dose of 50 mg/day. The dose will be increased weekly by 50 mg as tolerated to achieve a target dose of 200 mg/day. Patients will be treated for 12 months with thalidomide.
  Other Names: Thalomid™
  Arms: Auto transplants plus Therapy
Drug: Dexamethasone — Patients will receive dexamethasone at a dose of 40 mg per day during Days 1-4 of each month for 12 months. The first dose of dexamethasone to be given the same day the patient starts thalidomide.
  Other Names: Decadron, DexPak
  Arms: Auto transplants plus Therapy
Behavioral: Observation — One year of observation post-transplants.
  Arms: Auto and Allo transplants; Auto transplants

SUMMARY:
The study is designed as a Phase III, multi-center trial of tandem autologous transplants versus the strategy of autologous followed by Human Leukocyte Antigen (HLA)-matched sibling non-myeloablative allogeneic transplant. Study subjects will be biologically assigned to the appropriate arm depending on the availability of an HLA-matched sibling. There is a nested randomized phase III trial of observation versus maintenance therapy following the second autologous transplant for patients on the tandem autologous transplant arm.

DETAILED DESCRIPTION:
Multiple myeloma (MM), characterized by malignant plasma cell proliferation, bone destruction, and immunodeficiency, is a disease with a median age at diagnosis of approximately 65 years. It is responsible for about 1 percent of all cancer-related deaths in Western Countries. Conventional treatments with chemotherapy and radiation therapy are non-curative but improve quality of life and duration of survival. Attempts to cure myeloma through high-dose therapy followed by autografting or allografting have largely failed due to a combination of relapsed disease or transplant related mortality (TRM). High-dose therapy with autologous transplantation is safe and has low TRM (less than 5%), but is associated with a continuing and nearly universal risk of disease progression and relapse. Even so, autologous transplantation is superior to continued conventional chemotherapy. Recent data indicate that tandem autologous transplants are superior to a single procedure. Even with this approach, patients remain at risk of relapse and additional approaches are needed.

DESIGN NARRATIVE:

The overall study design is that of biologic assignment, based on the availability of an HLA-matched sibling, to one of two treatment strategies for MM patients. Patients without an HLA-matched sibling will undergo tandem autologous transplants. Patients with an HLA-matched sibling will undergo an autologous transplant followed by a non-myeloablative allogeneic transplant. In addition, the tandem autologous transplant recipients will be randomized to either observation or one year of maintenance therapy to begin following the second autologous transplant. The large number of MM patients without an HLA-matched sibling enables us to evaluate the role of maintenance therapy following tandem autologous transplants.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the Durie and Salmon criteria for initial diagnosis of MM
* Stage II or III MM at diagnosis or anytime thereafter
* Symptomatic MM requiring treatment at diagnosis or anytime thereafter
* Received at least three cycles of initial systemic therapy and are within 2-10 months of initiation of the initial therapy (this time frame excludes the time for mobilization therapy)
* If receiving chemotherapy-based mobilization regimens, must be able to receive high-dose melphalan between 2 and 8 weeks after the initiation of mobilization therapy whether delivered at the transplant center or at a referring center
* Adequate organ function as measured by:

  1. Cardiac: Left ventricular ejection fraction at rest greater than 40%
  2. Hepatic: Bilirubin less than 2 times the upper limit of normal and alanine transaminase (ALT) and aspartate transaminase (AST) less than 3 times the upper limit of normal
  3. Renal: Creatinine clearance greater than 40 ml/min (measured or calculated/estimated)
  4. Pulmonary: Carbon monoxide diffusion (DLCO), Volume forcibly exhaled in one second (FEV1), and Forced Vital Capacity (FVC) greater than 50% of predicted value (corrected for hemoglobin), or O2 saturation greater than 92% of room air
* An adequate autologous graft defined as a cryopreserved PBSC graft containing at least 4.0 x 106 CD34+ cells/kg patient weight; if prior to enrollment it is known that a patient will be on the auto-allo arm (i.e., a consenting, eligible HLA-matched sibling donor is available), the required autograft must contain at least 2.0 x 10^6 CD34+ cells/kg patient weight; the graft may not be CD34+ selected or otherwise manipulated to remove tumor or other cells; the graft can be collected at the transplanting institution or by a referring center; for patients without an HLA-matched sibling donor, the autograft must be stored so that there are two products each containing at least 2 x 10^6 CD34+ cells/kg patient weight

Exclusion Criteria:

* Never advanced beyond Stage I MM since diagnosis
* Non-secretory MM (absence of a monoclonal protein [M protein] in serum as measured by electrophoresis and immunofixation and the absence of Bence Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques)
* Plasma cell leukemia
* Karnofsky performance score less than 70%, unless approved by the Medical Monitor or one of the Protocol Chairs
* Uncontrolled hypertension
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms)
* Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the Medical Monitor or one of the Protocol Chairs; cancer treated with curative intent more than 5 years previously will be allowed
* Pregnant or breastfeeding
* Seropositive for the human immunodeficiency virus (HIV)
* Unwilling to use contraceptive techniques during and for 12 months following treatment
* Prior allograft or prior autograft
* Received mid-intensity melphalan (more than 50 mg IV) as part of prior therapy
* Prior organ transplant requiring immunosuppressive therapy

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2003-12; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (36):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope Samaritan, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Scripps Clinic/Green Hospital, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - BMT Group of Georgia/Northside Hospital, Atlanta, Georgia
  - Loyola University, Maywood, Illinois
  - IBMT (Indiana Blood and Marrow Transplant) at St Francis Franciscan Health, Indianapolis, Indiana
  - Wichita CCOP, Wichita, Kansas
  - Tufts - New England Medical Center, Boston, Massachusetts
  - DFCI/Brigham & Women's, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University (A), Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase - Temple University - BMT Program, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas/MD Anderson Cancer Research Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Utah BMT/Univ of Utah Med School, Salt Lake City, Utah
  - Virginia Commonwealth University MCV Hospitals, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Hospitals & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Krishnan A, Pasquini MC, Logan B, Stadtmauer EA, Vesole DH, Alyea E 3rd, Antin JH, Comenzo R, Goodman S, Hari P, Laport G, Qazilbash MH, Rowley S, Sahebi F, Somlo G, Vogl DT, Weisdorf D, Ewell M, Wu J, Geller NL, Horowitz MM, Giralt S, Maloney DG; Blood Marrow Transplant Clinical Trials Network (BMT CTN). Autologous haemopoietic stem-cell transplantation followed by allogeneic or autologous haemopoietic stem-cell transplantation in patients with multiple myeloma (BMT CTN 0102): a phase 3 biological assignment trial. Lancet Oncol. 2011 Dec;12(13):1195-203. doi: 10.1016/S1470-2045(11)70243-1. Epub 2011 Sep 29. PMID 21962393
- [Result] Logan B, Leifer E, Bredeson C, Horowitz M, Ewell M, Carter S, Geller N. Use of biological assignment in hematopoietic stem cell transplantation clinical trials. Clin Trials. 2008;5(6):607-16. doi: 10.1177/1740774508098326. PMID 19029209
- [Derived] Giralt S, Costa LJ, Maloney D, Krishnan A, Fei M, Antin JH, Brunstein C, Geller N, Goodman S, Hari P, Logan B, Lowsky R, Qazilbash MH, Sahebi F, Somlo G, Rowley S, Vogl DT, Vesole DH, Pasquini M, Stadtmauer E. Tandem Autologous-Autologous versus Autologous-Allogeneic Hematopoietic Stem Cell Transplant for Patients with Multiple Myeloma: Long-Term Follow-Up Results from the Blood and Marrow Transplant Clinical Trials Network 0102 Trial. Biol Blood Marrow Transplant. 2020 Apr;26(4):798-804. doi: 10.1016/j.bbmt.2019.11.018. Epub 2019 Nov 19. PMID 31756536
- Available data/document: Individual Participant Data Set: BMT CTN-0102 — http://biolincc.nhlbi.nih.gov/studies/bmtctn0102/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local Institutional Review Board (IRB) approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol: BMT CTN-0102 — http://biolincc.nhlbi.nih.gov/studies/bmtctn0102/
- Available data/document: Study Forms: BMT CTN-0102 — http://biolincc.nhlbi.nih.gov/studies/bmtctn0102/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between December 2003 and March 2007 from 37 different transplant centers.
Groups:
- Auto-Auto Standard Risk: Tandem autologous transplant plus thalidomide/dexamethasone (Thal-Dex) or observation (Obs) for standard risk patients PFS and OS did not differ between the Thal-Dex and the Obs arms and were thus pooled for analysis.
- Auto-Allo Standard Risk: Autologous transplant plus non-myeloablative allogeneic transplant for standard risk patients
- Auto-Auto High Risk: Tandem autologous transplant plus thalidomide/dexamethasone (Thal-Dex) or observation (Obs) for high risk patients
  PFS and OS did not differ between the Thal-Dex and the Obs arms and were thus pooled for analysis.
- Auto-Allo High Risk: Autologous transplant plus non-myeloablative allogeneic transplant for high risk patients
Period: Overall Study
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk
Started | 436 | 189 | 48 | 37
Completed | 178 (Participants that were alive and free of disease progression at the end of follow-up (3 years)) | 71 (Participants that were alive and free of disease progression at the end of follow-up (3 years)) | 14 (Participants that were alive and free of disease progression at the end of follow-up (3 years)) | 13 (Participants that were alive and free of disease progression at the end of follow-up (3 years))
Not Completed | 258 | 118 | 34 | 24

BASELINE CHARACTERISTICS:
Population: Analysis is based on intention-to-treat data. Primary analysis of the clinical trial focused on patients meeting protocol criteria of standard risk multiple myeloma.
Groups:
- Total: Total of all reporting groups
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk | Total
Number analyzed (Participants) | 436 | 189 | 48 | 37 | 710
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [22 to 70] | 53 [29 to 68] | 57 [32 to 70] | 51 [32 to 66] | 53.2 [22 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 78 | 21 | 16 | 291
  Male | 260 | 111 | 27 | 21 | 419
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 77 | 18 | 8 | 3 | 106
  Caucasian | 335 | 161 | 38 | 33 | 567
  Other | 24 | 10 | 2 | 1 | 37
Karnofsky Performance score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    100 - 90 | 344 | 148 | 27 | 26 | 545
    < 90 | 92 | 41 | 21 | 11 | 165
β-2 Microglobulin [Median (Full Range); unit: mg/L] | 2.0 [0.004 to 4.0] | 2.0 [0.9 to 4.0] | 4.4 [0.9 to 9.8] | 3.7 [1.2 to 6.6] | 3.025 [0.004 to 9.8]
Durie-Salmon [Number; unit: participants] — The Durie and Salmon classification uses three multiple myeloma stages. Stage I has all of the following: Hemoglobin greater than 10 g/dL, Serum calcium less than 12 mg/dL, Normal bone structure or solitary plasmacytoma on radiographs, and Low M component. Stage II does not fit either Stage I or Stage III. Stage III has one or more of the following: Hemoglobin less than 8.5 g/dL, Serum calcium greater than 12 mg/dL, Advanced lytic bone lesions, and/or Hyper M component.
  participants
    Stages I-II | 142 | 59 | 10 | 9 | 220
    Stage III | 294 | 130 | 38 | 28 | 490
Interval from diagnosis to transplantation [Median (Full Range); unit: months] | 7 [3 to 55] | 7 [4 to 35] | 7 [5 to 22] | 7 [3 to 38] | 7 [3 to 55]
Disease status [Number; unit: participants] — Disease status at time of first autologous transplantation represents the results from initial multiple myeloma therapy received prior to trial enrollment: Complete Response (CR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD)
  participants
    CR | 41 | 24 | 1 | 3 | 69
    Near CR | 65 | 22 | 1 | 2 | 90
    Very Good PR | 79 | 32 | 1 | 7 | 119
    PR | 158 | 76 | 21 | 14 | 269
    MR | 31 | 17 | 10 | 3 | 61
    SD | 21 | 6 | 6 | 4 | 37
    Not Evaluable | 30 | 12 | 8 | 4 | 54
    Unknown | 11 | 0 | 0 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Patients are considered a failure for this endpoint if they die or if they progress or relapse.
Time Frame: Year 3
Population: Patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Auto-Auto Standard Risk: Tandem autologous transplant plus thalidomide/dexamethasone or observation for standard risk patients
- Auto-Auto High Risk: Tandem autologous transplant plus thalidomide/dexamethasone or observation for high risk patients
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk
Number analyzed (Participants) | 366 | 156 | 31 | 29
percentage of patients | 46 [42 to 51] | 43 [36 to 51] | 33 [22 to 50] | 40 [27 to 60]

2. Secondary Outcome: Overall Survival (OS) for Standard Risk
Description: The event is death from any cause, patients alive at the time of last observation are considered censored.
Time Frame: Years 1, 2, and 3
Population: Patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk
Number analyzed (Participants) | 366 | 156
percentage of patients
  1 year | 95 [93 to 97] | 91 [87 to 95]
  2 years | 89 [86 to 92] | 85 [80 to 91]
  3 years | 80 [77 to 84] | 77 [72 to 84]

3. Secondary Outcome: Overall Survival (OS) for High Risk
Description: The event is death from any cause, patients alive at the time of last observation are considered censored.
Time Frame: Year 3
Population: Patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Auto-Auto High Risk | Auto-Allo High Risk
Number analyzed (Participants) | 31 | 29
percentage of participants | 67 [54 to 82] | 59 [45 to 78]

4. Secondary Outcome: Cumulative Incidence of Progression/Relapse
Description: Patients are considered experiencing an event when they progress. Deaths without progression are considered as a competing risk. Patients initiating non-protocol anti-myeloma therapy are considered to have progressed on this protocol.
Time Frame: Year 3
Population: Patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk
Number analyzed (Participants) | 366 | 156 | 31 | 29
percentage of patients | 50 [46 to 55] | 46 [39 to 54] | 57 [42 to 71] | 38 [22 to 54]

5. Secondary Outcome: Cumulative Incidence of Treatment Related Mortality (TRM)
Description: TRM is defined as death occurring in a patient from causes other than relapse or progression.
Time Frame: Year 3
Population: Patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk
Number analyzed (Participants) | 366 | 156 | 31 | 29
percentage of participants | 4 [2 to 5] | 11 [7 to 16] | 11 [2 to 19] | 22 [8 to 35]

6. Secondary Outcome: Interval From First to Second Transplantation
Description: Upon recovery from the first autograft, but at least 60 days (preferably between 60-120 days) after the first autograft, patients will receive a second transplant according to treatment assignments.
Time Frame: Year 1
Population: Patients that completed second transplant
Measure: Median (Full Range); unit: days
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk
Number analyzed (Participants) | 366 | 156 | 31 | 29
days | 98 [58 to 193] | 105 [61 to 262] | 101 [63 to 155] | 111 [61 to 155]

7. Secondary Outcome: Incidences of Graft Versus Host Disease (GVHD)
Description: Incidence and severity of GVHD will be scored according to the BMT clinical trials network Manual of Procedures.
Time Frame: Day 100
Population: GVHD was only assessed on the Auto-Allo arm for standard risk patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Auto-Allo Standard Risk
Number analyzed (Participants) | 156
percentage of patients
  Grades II-IV | 26 [19 to 33]
  Grades III-IV | 9 [4 to 14]

8. Secondary Outcome: Incidences of Chronic GVHD
Description: Incidence and severity of chronic GVHD will be scored according to the BMT clinical trials network Manual of Procedures.
Time Frame: Years 1 and 2
Population: GVHD was only assessed on the Auto-Allo arm for standard risk patients that completed second transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Auto-Allo Standard Risk
Number analyzed (Participants) | 156
percentage of patients
  1 year | 47 [39 to 56]
  2 years | 54 [46 to 63]

ADVERSE EVENTS:
Time Frame: 3-years post-first transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected adverse events were required to be reported through the adverse event system per protocol.
Arm/Group | Auto-Auto Standard Risk | Auto-Allo Standard Risk | Auto-Auto High Risk | Auto-Allo High Risk
Serious Adverse Events (participants affected / at risk) | 15/436 | 10/189 | 2/48 | 5/37
Other Adverse Events (participants affected / at risk) | 1/436 | 1/189 | 0/48 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Auto-Auto Standard Risk (N=436) | Auto-Allo Standard Risk (N=189) | Auto-Auto High Risk (N=48) | Auto-Allo High Risk (N=37)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Accidental death (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Engraftment syndrome (Immune system disorders) | 1 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral cardiomyopathy (Infections and infestations) | 1 | 0 | 0 | 0
Delayed engraftment (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fever (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Gallbladder operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than .2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-Auto Standard Risk (N=436) | Auto-Allo Standard Risk (N=189) | Auto-Auto High Risk (N=48) | Auto-Allo High Risk (N=37)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2006-05-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT00075829/Prot_SAP_ICF_000.pdf